CLINICAL TRIAL: NCT06958705
Title: Study of the Efficacy and Safety of Venetoclax as Consolidation to Achieve Fix-Duration Treatment in CLL Patients Treated With BTK Inhibitor Monotherapy
Brief Title: Venetoclax as Consolidation in CLL Patients Treated With BTK Inhibitor Monotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-1147
Record Dates: First submitted 2025-04-08; First posted 2025-05-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-04

CONDITIONS: Chronic Lymphocytic Leukemia (CLL) / Small Lymphocytic Lymphoma (SLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; zanubrutinib; acalabrutinib; orelabrutinib

STUDY DESIGN:
Intervention Model Description: Patients will be treated with the BTK inhibitor plus full-dose venetoclax for 12 cycles after a standard 5-week dose ramp-up. Peripheral blood and bone marrow MRD status will be evaluated during and after the treatment. After the completion of combination therapy, patients will stop both BTK inhibitor and venetoclax and be followed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CLL/SLL patients on ibrutinib monotherapy for ≥ 6 months (Experimental)
  Interventions: Drug: Venetoclax combined with Ibrutinib
- CLL/SLL patients on zanubrutinib monotherapy for ≥ 6 months (Experimental)
  Interventions: Drug: Venetoclax combined with Zanubrutinib
- CLL/SLL patients on acalabrutinib monotherapy for ≥ 6 months (Experimental)
  Interventions: Drug: Venetoclax combined with Acalabrutinib
- CLL/SLL patients on orelabrutinib monotherapy for ≥ 6 months (Experimental)
  Interventions: Drug: Venetoclax combined with Orelabrutinib

INTERVENTIONS:
Drug: Venetoclax combined with Ibrutinib — All Patients will be treated with venetoclax for 12 cycles after a standard 5-week dose ramp-up, as an add-on to the primary using ibrutinib. After the completion of combination therapy, patients will stop both the ibrutinib and venetoclax then be followed.
  Each cycle is 28 days. At the start of cycle 0, patients will start venetoclax by 20mg-50mg-100mg-200mg daily in a weekly dose escalation way. The combination of full dose venetoclax (400mg) and ibrutinib will continue for an additional 12 cycles. Venetoclax and ibrutinib will be continued until the completion of cycle 12, start of new CLL-directed therapies, disease progression or unacceptable toxicities, depending on which comes first.
  Ibrutinib is intended to be admistratered orally 420mg once daily.
  Arms: CLL/SLL patients on ibrutinib monotherapy for ≥ 6 months
Drug: Venetoclax combined with Zanubrutinib — All Patients will be treated with venetoclax for 12 cycles after a standard 5-week dose ramp-up, as an add-on to the primary using zanubrutinib. After the completion of combination therapy, patients will stop both the zanubrutinib and venetoclax then be followed.
  Each cycle is 28 days. At the start of cycle 0, patients will start venetoclax by 20mg-50mg-100mg-200mg daily in a weekly dose escalation way. The combination of full dose venetoclax (400mg) and zanubrutinib will continue for an additional 12 cycles. Venetoclax and zanubrutinib will be continued until the completion of cycle 12, start of new CLL-directed therapies, disease progression or unacceptable toxicities, depending on which comes first.
  Zanubrutinib is intended to be admistratered orally 160mg twice daily.
  Arms: CLL/SLL patients on zanubrutinib monotherapy for ≥ 6 months
Drug: Venetoclax combined with Acalabrutinib — All Patients will be treated with venetoclax for 12 cycles after a standard 5-week dose ramp-up, as an add-on to the primary using acalabrutinib. After the completion of combination therapy, patients will stop both the acalabrutinib and venetoclax then be followed.
  Each cycle is 28 days. At the start of cycle 0, patients will start venetoclax by 20mg-50mg-100mg-200mg daily in a weekly dose escalation way. The combination of full dose venetoclax (400mg) and acalabrutinib will continue for an additional 12 cycles. Venetoclax and acalabrutinib will be continued until the completion of cycle 12, start of new CLL-directed therapies, disease progression or unacceptable toxicities, depending on which comes first.
  Acalabrutinib is intended to be admistratered orally 100mg twice daily.
  Arms: CLL/SLL patients on acalabrutinib monotherapy for ≥ 6 months
Drug: Venetoclax combined with Orelabrutinib — All Patients will be treated with venetoclax for 12 cycles after a standard 5-week dose ramp-up, as an add-on to the primary using orelabrutinib. After the completion of combination therapy, patients will stop both the orelabrutinib and venetoclax then be followed.
  Each cycle is 28 days. At the start of cycle 0, patients will start venetoclax by 20mg-50mg-100mg-200mg daily in a weekly dose escalation way. The combination of full dose venetoclax (400mg) and orelabrutinib will continue for an additional 12 cycles. Venetoclax and orelabrutinib will be continued until the completion of cycle 12, start of new CLL-directed therapies, disease progression or unacceptable toxicities, depending on which comes first.
  Orelabrutinib is intended to be admistratered orally 150mg once daily.
  Arms: CLL/SLL patients on orelabrutinib monotherapy for ≥ 6 months

SUMMARY:
This is an open-label, multicenter, phase 2, non-randomized study aiming to study the efficacy and safety of fixed-duration venetoclax consolidation in CLL patients who are on BTK inhibitor monotherapy. Patients who are on BTK inhibitor monotherapy for ≥ 6 months and still responsive are included. The study includes patients who are treatment-naive before taking BTK inhibitors. Patients will be treated with the BTK inhibitor plus full-dose venetoclax for 12 cycles after a standard 5-week dose ramp-up. Peripheral blood and bone marrow MRD status will be evaluated during and after the treatment. After the completion of combination therapy, patients will stop both BTK inhibitor and venetoclax and be followed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18-80 years-old.
* 2. Patients must have a diagnosis of CLL/SLL.
* 3. Detectable MRD by flow cytometry (10^-4 sensitivity) in the peripheral blood.
* 4. Patients who are on BTK inhibitor monotherapy for more than 6 months. This study includes patients who are taking one of the following BTK inhibitors: ibrutinib, zanubrutinib, orelabrutinib, and acalabrutinib.
* 5. Patients need to have a response of at least PR (CR/PR) to BTK inhibitor monotherapy.
* 6. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* 7. Patients must have adequate renal and hepatic function:
* Serum bilirubin ≤ 1.5 × upper limit of normal (ULN) or ≤ 3 × ULN for patients with Gilbert's disease;
* Serum creatinine clearance of ≥ 50 ml/min (calculated or measured);
* ALT and AST ≤ 3.0 × ULN, unless clearly due to disease involvement.
* 8. Adequate bone marrow function:
* Platelet count of greater than 50,000/µl, with no platelet transfusion in prior 2 weeks;
* ANC ≥ 1000/µl in the absence of growth factor support unless due to compromised bone marrow production from CLL, indicated by ≥ 80% CLL in marrow;
* Hemoglobin ≥ 8g/dL.
* 9. Adequate cardiac function, as assessed by:
* Absence of uncontrolled cardiac arrhythmia;
* Echocardiogram demonstrating LVEF ≥ 35%;
* NYHA functional class ≤ 2.
* 10. Ability to provide informed consent and adhere to the required follow-up.

Exclusion Criteria:

* 1. Richter transformation.
* 2. Active malignancy requiring systemic therapy, other than CLL, with the exception of: adequately treated in situ carcinoma of the cervix uteri; adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin; previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
* 3. Major surgery, radiotherapy, chemotherapy, biologic therapy, immunotherapy, experimental therapy within 3 weeks prior to the first dose of the study drug.
* 4. Grade 3 or 4 hemorrhage within the past 3 weeks.
* 5. Uncontrolled active infections (viral, bacterial, and fungal).
* 6. Females who are pregnant or lactating.
* 7. Known HIV positive.
* 8. Active hepatitis B infection (defined as the presence of detectable HBV DNA or HBe antigen). Patients who are HBsAg positive or HBcAb positive are eligible, provided HBV DNA is negative. These patients must have monthly monitoring of HBV DNA for the duration of the study.
* 9. Active hepatitis C, defined by the detection of hepatitis C RNA in plasma by PCR.
* 10. Active, uncontrolled autoimmune phenomenon (autoimmune hemolytic anemia or immune thrombocytopenia) requiring steroid therapy > 20 mg prednisone daily or equivalent, within 7 days of starting venetoclax.
* 11. Received other therapeutic agents for CLL/SLL during BTK inhibitor treatment prior to enrollment.
* 12. Concurrent use of warfarin or equivalent vitamin K inhibitor or other oral anticoagulant treatment.
* 13. Received strong CYP3A inhibitors or strong CYP3A inducers within 7 days of starting venetoclax.
* 14. Consuming grapefruit, grapefruit products, Seville oranges, or star fruit within 7 days of starting venetoclax.
* 15. Prior treatment with venetoclax or other Bcl-2 inhibitor.
* 16. Malabsorption syndrome or other condition that precludes enteral route of administration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of BM-uMRD after completion of combination therapy (Day 1 of Cycle 16) | On Day 1 of Cycle 16 (each cycle is 28 days)
  Rate of BM-uMRD is defined by negative MRD in the bone marrow by flow cytometry at a sensitivity of 10^-4. The Clopper Pearson method is used to estimate the 95% two-sided confidence interval (CI) of the rate of BM-uMRD.

SECONDARY OUTCOMES:
Rate of undetected peripheral blood MRD by flow cytometry | On screening, Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 10, Day 1 of Cycle 16, Day 1 of Cycle 20, Day 1 of Cycle 24, Day 1 of Cycle 28 and Day 1 of Cycle 34 (each cycle is 28 days)
  Rate of undetected peripheral blood MRD is defined by negative MRD in the peripheral blood by flow cytometry at a sensitivity of 10^-4.
Rate of complete response (CR) | On Day 1 of Cycle 7, Day 1 of Cycle 16, Day 1 of Cycle 22, and Day 1 of Cycle 28 (each cycle is 28 days)
  CR is defined by the 2018 IWCLL criteria. Enhanced contrast CT combined with bone marrow examination will be performed to determine if a patient achieve CR.
Progression-free survival (PFS) | From the first dose of venetoclax until the date of progression or date of death from any cause, whichever came first, assessed up to 112 months
  PFS is defined as the time from the first dose of venetoclax to progression, or death due to any cause, whichever occurs first. For subjects without progression, relapse, or death at the time of analysis, EFS will be censored at the last assessment date.
Overall survival (OS) | From the first dose of venetoclax until the date of death from any cause, assessed up to 112 months
  OS is defined as the time from the first dose of venetoclax to death due to any cause. Subjects who remain alive at the time of analysis will be censored at the last known alive date of the subject.
Time to next treatment (TTNT) | From the first dose of venetoclax to the next CLL-directed therapies due to progression, assessed up to 112 months
  TTNT is defined as the time from the first dose of venetoclax to the next CLL-directed therapies.
Adverse Events | From screening to 30 days after the end of cycle 12 (each cycle is 28 days)
  All treatment-emergent AEs will be included in the analysis. For each AE, the number and percentage of subjects who experience at least one occurrence of the given event will be summarized. The number and percent of subjects with TEAEs will be summarized according to intensity (CTCAE, v5) or IWCLL for hematologic toxicity, and drug relationship, as well as categorized by system organ class and preferred term. Summaries, listings, datasets, or subject narratives may be provided, as appropriate, for those subjects who die, who discontinue treatment due to an AE, or who experience a severe AE or a SAE.

OTHER OUTCOMES:
MRD relapse | From the date of MRD negativity to the date of MRD positivity or the occurrence of increase of MRD ≥ 1 log10 between any 2 positive samples measured in the same tissue, assessed up to 112 months
  MRD relapse is now defined as either: (1) conversion of MRD negativity to MRD positivity, independent of the MRD technique, or (2) increase of MRD ≥ 1 log10 between any 2 positive samples measured in the same tissue (PB or BM) in patients with MRD+ CLL.
Clearance of BTK C481S mutation | On Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 10, and Day 1 of Cycle 16 (each cycle is 28 days)
  Baseline BTK C418S mutation by droplet digital PCR will performed. Patients with detected baseline BTK C481S mutation will be re-evaluated at C4D1, C7D1, C10D1, and C16D1 to determine the effects of venetoclax on the clearance of BTK C481S mutation.
Occurance of laboratory or clinical TLS | From Day 1 of Cycle 0 to Day 28 of Cycle 0 (dose ramp-up phase)
  In the dose ramp-up phase, laboratory and clinical monitoring will be regularly performed to determine if TLS occur.
MRD level detected by NGS IG sequencing | On Day 1 of Cycle 0, Day 1 of Cycle 4, Day 1 of Cycle 7, Day 1 of Cycle 10, and Day 1 of Cycle 16 (each cycle is 28 days)
  Peripheral blood MRD by NGS of immunoglobulin (IG) will be evaluated at C0D1, C4D1, C7D1, C10D1, and C16D1. NGS of IG for determining bone marrow MRD status will be performed at C0D1, C7D1, and C16D1. At the timepoints, the correlation between MRD by flow cytometry and NGS MRD will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Haematology, the First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital, Nanjing, Jiangsu, China